CLINICAL TRIAL: NCT01810484
Title: Feasibility Study: Evaluation of the Ulthera® System in Combination With 70W Alma Pixel CO2 Fractional Ablative Laser for Improvement of Abdominal Striae
Brief Title: Feasibility Study: Evaluation of the Treatment of Striae Using Ultherapy® in Combination With Laser Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-133
Record Dates: First submitted 2013-03-08; First posted 2013-03-13 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2015-01

CONDITIONS: Scars; Striae
Keywords: Ulthera® System; Ultherapy® Treatment; Ulthera, Inc.; Ultrasound treatment for skin
MeSH Terms: conditions — Cicatrix; Striae Distensae

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): The abdominal region will be divided into 3 treatment areas: Treatment Area A, B and C.
  Treatment Area A will be treated with Ultherapy® treatment only; Treatment Area B will be treated with Ultherapy® treatment and CO2 laser treatment; Treatment Area C will be treated with CO2 laser treatment only
  Interventions: Device: Ultherapy® treatment only; Device: Ultherapy® treatment and CO2 laser treatment; Device: CO2 Laser treatment only
- Group 2 (Active Comparator): The abdominal region will be divided into 3 treatment areas: Treatment Area A, B and C.
  Treatment Area A will be treated with Ultherapy® treatment and CO2 laser treatment; Treatment Area B will be treated with CO2 laser treatment only; Treatment Area C will be treated with Ultherapy® treatment only
  Interventions: Device: Ultherapy® treatment only; Device: Ultherapy® treatment and CO2 laser treatment; Device: CO2 Laser treatment only
- Group 3 (Active Comparator): The abdominal region will be divided into 3 treatment areas: Treatment Area A, B and C.
  Treatment Area A will be treated with CO2 laser treatment only; Treatment Area B will be treated with Ultherapy® treatment only; Treatment Area C will be treated with Ultherapy® treatment and CO2 laser treatment
  Interventions: Device: Ultherapy® treatment only; Device: Ultherapy® treatment and CO2 laser treatment; Device: CO2 Laser treatment only

INTERVENTIONS:
Device: Ultherapy® treatment only — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ulthera® System treatment
Device: Ultherapy® treatment and CO2 laser treatment — Ultherapy® treatment: Focused ultrasound energy delivered below the surface of the skin;
  CO2 Laser: Fractionated energy delivered to the surface of the skin for ablative and thermal injury to the skin layers for resurfacing the skin.
  Other Names: Ulthera® System treatment; CO2 Fractional Ablative Laser teatment
Device: CO2 Laser treatment only — CO2 Laser: Fractionated energy delivered to the surface of the skin for ablative and thermal injury to the skin layers for resurfacing the skin.
  Other Names: CO2 Fractional Ablative Laser teatment

SUMMARY:
Up to 20 subjects will be enrolled. Enrolled subjects will receive one of three study treatments in the abdominal region: Ultherapy® only, Ultherapy® and CO2 laser treatment, or CO2 laser treatment only. Follow-up visit will occur at 14, 90 and 180 days post-treatment. Study images will be obtained pre-treatment, approximately 30 minutes post-treatment, and at each follow-up visit.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blinded, pilot clinical trial to evaluate the use of the Ulthera® System in combination with the 70W Alma Pixel CO2 laser for efficacious results in the treatment of abdominal striae rubra and striae alba. Subjects will be randomized to one of three treatment groups. Study personnel conducting efficacy measures will be blinded to the assigned treatment groups.

Changes from baseline in overall skin texture and appearance of abdominal striae will be assessed at study follow-up visits. 2D images, 3D images and patient satisfaction questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 21 to 65 years.
* Subject in good health.
* Fitzpatrick skin classification type 1-5.
* Striae rubra and alba on the abdomen.
* Understands and accepts the obligation not to undergo any other procedures in the area(s) to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Absence of physical or psychological conditions unacceptable to the investigator.
* Willingness and ability to provide written consent for study-required photography and adherence to photography requirements .
* Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1 and be willing and able to use an acceptable method of birth control during the study

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Current bacterial or viral infection in the area to be treated.
* Severe solar elastosis.
* Significant scarring or burns in area(s) to be treated.
* Prior radiation therapy in the area(s) to be treated.
* Open wounds or lesions in the area(s) to be treated.
* History of keloid or hypertrophic scarring
* History of irregular pigmentation of the skin, Lichens Planus, Vitiligo or Psoriasis in the treatment area that in the investigators opinion, would put the subject at unnecessary risk.
* Inability to understand the protocol or to give informed consent.
* Microdermabrasion, or prescription level glycolic acid treatments to the intended treatment area(s) within two weeks prior to study participation or during the study.
* History of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
* Subjects who anticipate the need for surgery or overnight hospitalization during the study.
* Subjects who, in the investigator's opinion, have a history of poor cooperation,noncompliance with medical treatment, or unreliability.
* Concurrent enrollment in any study involving the use of investigational devices or drugs.
* Current smoker or history of smoking in the last five years.
* History of prior abdominal Suction Assisted Lipectomy or Abdominoplasty.
* History of prior Massive Weight Loss
* History of using the following prescription medications:

  1. Accutane or other systemic retinoids within the past 12 months;
  2. Antiplatelet agents / Anticoagulants (Coumadin, Heparin, Plavix);
  3. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing informed consent.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in overall skin texture and appearance of abdominal striae | 90-days post-treatment
  A masked, qualitative assessment of change from baseline in the areas treated based a review of 2D images obtained at baseline and 90 days post-treatment.

SECONDARY OUTCOMES:
90 Day Patient Satisfaction | 90 Days post-treatment
  Based on completion of Patient Satisfaction Questionnaires
180 Day Patient Satisfaction | 180 Days post-treatment
  Based on completion of Patient Satisfaction Questionnaires
Change from baseline in overall aesthetic appearance of abdominal striae at 90 days | 90 Days post-treatment
  Assessment of change in overall aesthetic appearance of abdominal striae from baseline to 90 days post-treatment based on review of pretreatment and 90 day post-treatment 2D images and a live assessment of the treatment area
Change from baseline in overall aesthetic appearance of abdominal striae at 180 days | 180 Days post-treatment
  Assessment of change in overall aesthetic appearance of abdominal striae from baseline to 180 days post-treatment based on review of pretreatment and 180 day post-treatment 2D images and a live assessment of the treatment area
Change from baseline in skin striae texture and depth at 90 Days | 90 Days post-treatment
  Quantitative analysis will be completed comparing 3D images obtained at baseline to 3D images obtained at 90 days post-treatment.
Change from baseline in skin striae texture and depth at 180 Days | 180 Days post-treatment
  Quantitative analysis will be completed comparing 3D images obtained at baseline to 3D images obtained at 180 days post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Zapiach, MD, Principal Investigator — Art Plastic Surgery
Locations (2):
- United States (2):
  - Art Plastic Surgery, Paramus, New Jersey
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina